CLINICAL TRIAL: NCT00210236
Title: Surgical Resection With or Without Axillary Lymph Node Excision in Treating Menopausal Women With Infiltrative Breast Cancer Smaller Than 10 mm
Brief Title: Surgical Breast Resection With or Without Axillary Lymph Node Excision in Treating Women With Breast Cancer
Acronym: AXIL95
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB1995-28
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Breast neoplasms; Local recurrence; Survival; Surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy

ARMS (2):
- Conventional surgery WITH Axillary Lymph Node Excision (Experimental): Tumorectomy or mastectomy, WITH Axillary Lymph Node Excision
  Interventions: Procedure: Conventional surgery WITH Axillary Lymph Node Excision
- Conventional surgery WITHOUT Axillary Lymph Node Excision (Active Comparator): Tumorectomy or mastectomy, WITHOUT Axillary Lymph Node Excision
  Interventions: Procedure: Conventional surgery WITHOUT Axillary Lymph Node Excision

INTERVENTIONS:
Procedure: Conventional surgery WITHOUT Axillary Lymph Node Excision — Tumorectomy or mastectomy, WITHOUT Axillary Lymph Node Excision
  Arms: Conventional surgery WITHOUT Axillary Lymph Node Excision
Procedure: Conventional surgery WITH Axillary Lymph Node Excision
  Other Names: Tumorectomy or mastectomy, WITH Axillary Lymph Node Excision
  Arms: Conventional surgery WITH Axillary Lymph Node Excision

SUMMARY:
This randomized phase III trial is studying surgery and axillary lymph node dissection to evaluate if systematic Axillary Lymph Node Excision can be avoided in locoregional treatment for operable breast cancer smaller than 10 mm among menopausal women older than 50

DETAILED DESCRIPTION:
Phase III randomized multicenter equivalence trial evaluating the role of Axillary Lymph Node Excision.

Primary aim is to assess if it is possible to avoid routine Axillary Lymph Node Excision during the initial treatment of breast cancers smaller than 11 mm in women aged 50 and older without compromising survival? The primary endpoint is overall survival: the event considered will be death from any cause.

ELIGIBILITY:
Inclusion criteria:

Women, 50 year or more Menopausal women Breast cancer Macroscopic tumor size of 10 mm or less (measured during operation) No palpable axillary node ( N0)

Exclusion criteria:

Previous cancer history life expectancy < 10 years Metastasis

Ages: 50 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 625 (Actual)
Dates: Start 1995-09 (Actual); Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine AVRIL, MD, Principal Investigator — Institut Bergonié
Locations (14):
- France (14):
  - Centre Hospitalier Universitaire d'Agen, Agen
  - Centre Régional de Lutte Contre le Cancer d'Anger, Angers
  - Institut Bergonié - Centre Régional de Luttre Contre le Cancer de Bordeaux et du Sud Ouest, Bordeaux
  - Centre Régional de Luttre Contre le Cancer de Clermont Ferrand, Clermont-Ferrand
  - Centre Régional de Luttre Contre le Cancer de Dijon, Dijon
  - Centre Régional de Luttre Contre le Cancer de Lille, Lille
  - Centre Régional de Lutte Contre le Cancer de Lyon, Lyon
  - Centre Hospitalier Intercommunal de Marmande, Marmande
  - Centre Régional de Luttre Contre le Cancer de Montpellier, Montpellier
  - Clinique de la Source, Orléans
  - Centre Régional de Luttre Contre le Cancer de Nantes, Saint-Herblain
  - Centre Hospitalier Universitaire de Saint Nazaire, Saint-Nazaire
  - Centre Régional de Luttre Contre le Cancer de Strasbourg, Strasbourg
  - Centre Regional de Lutte Contre le Cancer de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Avril A, Le Bouedec G, Lorimier G, Classe JM, Tunon-de-Lara C, Giard S, MacGrogan G, Debled M, Mathoulin-Pelissier S, Mauriac L; AXIL95 Group. Phase III randomized equivalence trial of early breast cancer treatments with or without axillary clearance in post-menopausal patients results after 5 years of follow-up. Eur J Surg Oncol. 2011 Jul;37(7):563-70. doi: 10.1016/j.ejso.2011.04.008. Epub 2011 Jun 12. PMID 21665421

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional Surgery WITH Axillary Lymph Node Excision: Tumorectomy or mastectomy, WITH Axillary Lymph Node Excision
  Conventional surgery WITH Axillary Lymph Node Excision
Period: Overall Study
Arm/Group | Conventional Surgery WITH Axillary Lymph Node Excision | Conventional Surgery WITHOUT Axillary Lymph Node Excision
Started | 313 | 312
Completed | 313 | 312
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Surgery WITH Axillary Lymph Node Excision | Conventional Surgery WITHOUT Axillary Lymph Node Excision | Total
Number analyzed (Participants) | 313 | 312 | 625
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (7.2) | 62.9 (7.0) | 62.9 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 313 | 312 | 625
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 313 | 312 | 625

OUTCOME MEASURES:

1. Primary Outcome: Number of Deaths
Time Frame: Five years after surgery
Population: Per protocol population.
  The following patients were excluded from the PP population :
  * patients who did not satisfy eligibility criteria
  * patients who did receive the intervention as allocated by the randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Surgery WITH Axillary Lymph Node Excision | Conventional Surgery WITHOUT Axillary Lymph Node Excision
Number analyzed (Participants) | 310 | 297
Participants | 6 | 17
Statistical Analysis 1: Comparison: Conventional Surgery WITH Axillary Lymph Node Excision vs Conventional Surgery WITHOUT Axillary Lymph Node Excision; Test type: Equivalence — The two groups will be considered equivalent if the 5-year survival rate for group B (without lymph node dissection) is not less than 92%. This corresponds to hazard ratio (HR) of less than 1.6; p = 0.013, Log Rank; Hazard Ratio (HR) = 3.067, 95% CI 2-sided [1.4 to 6.7]

2. Secondary Outcome: Rate of Axillary Recurrence
Description: Proportion of participants with axiallary recurrence. Axillary (Regional) recurrence is defined as tumor recurrence in lymph nodes draining the primary tumor site, namely, nodes in the ipsilateral axilla, infraclavicular fossa, supraclavicular fossa and interpectoral area.
Time Frame: Five years after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Surgery WITH Axillary Lymph Node Excision | Conventional Surgery WITHOUT Axillary Lymph Node Excision
Number analyzed (Participants) | 310 | 297
Participants | 0 | 7

ADVERSE EVENTS:
Time Frame: 10 years
Description: Serious and non-serious adverse events were not collected.
Arm/Group | Conventional Surgery WITH Axillary Lymph Node Excision | Conventional Surgery WITHOUT Axillary Lymph Node Excision
All-Cause Mortality (participants affected / at risk) | 10/313 | 24/312
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes